CLINICAL TRIAL: NCT00491530
Title: A Year 2, Long-Term, Open-Label, Safety Extension Study of the Combination of ABT-335 and Statin Therapy for Subjects With Mixed Dyslipidemia
Brief Title: A Year 2, Safety Extension Study of the Combination of ABT-335 and Statin Therapy for Subjects With Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06-884
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Results first posted 2009-12-07 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Mixed Dyslipidemia
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; fenofibric acid; Rosuvastatin Calcium; Simvastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-335 + rosuvastatin calcium (Experimental)
  Interventions: Drug: ABT-335; Drug: rosuvastatin calcium
- ABT-335 + simvastatin (Experimental)
  Interventions: Drug: ABT-335; Drug: simvastatin
- ABT-335 + atorvastatin calcium (Experimental)
  Interventions: Drug: ABT-335; Drug: atorvastatin calcium

INTERVENTIONS:
Drug: ABT-335 — Oral coadministration of ABT-335 (135 mg) once daily, beginning in either the 12-week double-blind study or the previous 52-week open-label year 1 study and continuing in 52-week year 2 study
  Other Names: fenofibric acid
Drug: rosuvastatin calcium — Oral coadministration of rosuvastatin calcium (20 mg) once daily, beginning in either the 12-week double-blind study or the previous 52-week open-label year 1 study and continuing in 52-week year 2 study
  Other Names: Crestor
  Arms: ABT-335 + rosuvastatin calcium
Drug: simvastatin — Oral coadministration of simvastatin (40 mg) once daily, beginning in either the 12-week double-blind study or the previous 52-week open-label year 1 study and continuing in 52-week year 2 study
  Other Names: Zocor
  Arms: ABT-335 + simvastatin
Drug: atorvastatin calcium — Oral coadministration of atorvastatin calcium (40 mg) once daily, beginning in either the 12-week double-blind study or the previous 52-week open-label year 1 study and continuing in 52-week year 2 study
  Other Names: Lipitor
  Arms: ABT-335 + atorvastatin calcium

SUMMARY:
The objective of the study is to assess the continued safety of the daily coadministration of ABT-335 in combination with rosuvastatin calcium, simvastatin or atorvastatin calcium.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects who voluntarily sign the informed consent.
* Subject has successfully completed the treatment phase of the preceding open-label year 1 study.

Exclusion Criteria:

* Subject is using or will use investigational medications, except as approved by Abbott.
* Subject has prematurely discontinued his/her combination therapy administered in the preceding open-label year 1 study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Information Specialist, Abbott Park, Illinois, United States

REFERENCES:
- [Derived] Kipnes MS, Roth EM, Rhyne JM, Setze CM, Lele A, Kelly MT, Sleep DJ, Stolzenbach JC. Year two assessment of fenofibric acid and moderate-dose statin combination: a phase 3, open-label, extension study. Clin Drug Investig. 2010;30(1):51-61. doi: 10.2165/11319800-000000000-00000. PMID 19995098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had completed ABT-335/statin therapy in the preceding open-label year 1 study at a subset of sites were eligible for recruitment in this open-label year 2 extension study. Subjects continued to receive the treatment they had received in the preceding open-label year 1 study.
Groups:
- ABT-335 + 20 mg Rosuvastatin: Oral coadministration of ABT-335 (135 mg) + rosuvastatin (20 mg), once daily, for up to 116 weeks (if beginning in the 12-week double-blind study) or up to 104 weeks (if beginning in the previous 52-week open-label year 1 study) and continuing in 52-week year 2 study
- ABT-335 + 40 mg Simvastatin: Oral coadministration of ABT-335 (135 mg) + simvastatin (40 mg), once daily, for up to 116 weeks (if beginning in the 12-week double-blind study) or up to 104 weeks (if beginning in the previous 52-week open-label year 1 study) and continuing in 52-week year 2 study
- ABT-335 + 40 mg Atorvastatin: Oral coadministration of ABT-335 (135 mg) + atorvastatin (40 mg), once daily, for up to 116 weeks (if beginning in the 12-week double-blind study) or up to 104 weeks (if beginning in the previous 52-week open-label year 1 study) and continuing in 52-week year 2 study
Period: Overall Study
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Started | 174 | 50 | 86
Completed | 162 | 44 | 81
Not Completed | 12 | 6 | 5
Not completed — Adverse Event | 6 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Investigator Discretion | 0 | 1 | 0
Not completed — Patient Request | 0 | 1 | 0
Not completed — Use of Prohibited Medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin | Total
Number analyzed (Participants) | 174 | 50 | 86 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 138 | 40 | 68 | 246
  >=65 years | 36 | 10 | 18 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (10.71) | 55.3 (10.55) | 55.4 (10.94) | 55.8 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 29 | 42 | 148
  Male | 97 | 21 | 44 | 162
Region of Enrollment [Number; unit: participants]
  United States | 174 | 50 | 86 | 310

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Reporting Adverse Events During Combination Therapy in the Preceding Double-Blind Studies or in the Preceding Open-Label Year 1 Study or in This Open-Label Year 2 Study
Description: All serious and non-serious adverse events are reported from the time of combination study drug initiation until 30 days after discontinuation of study drug. Adverse events are unfavorable changes in health that occur in subjects during a clinical trial or within a specified period following a trial. Serious adverse events are those that result in death, require inpatient hospitalization or the prolongation of hospitalization, result in congenital anomaly/birth defect, or significant disability/incapacity or are life-threatening.
Time Frame: Anytime after initiation of combination therapy (in the preceding 12-week double-blind studies or in the preceding open-label year 1 study) up to 116 weeks, to within 30 days after the last dose of combination therapy.
Population: Subjects who took at least 1 dose of ABT-335 plus a statin in the preceding double-blind studies or preceding open-label year 1 study, and in this open-label year 2 study. All adverse events in the preceding studies or in this study occurring with exposure to combination therapy are summarized.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 174 | 50 | 86
percentage of participants | 94.8 | 90.0 | 97.7

2. Secondary Outcome: Median Percent Change in Triglycerides From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 triglycerides minus baseline triglycerides)/baseline triglycerides] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: Baseline to Week 104 (may include weeks in preceding double-blind studies [combination treatment arms], plus 52 weeks in preceding open-label year 1 study, and open-label year 2 study, up to 104 weeks)
Population: Subjects who took at least 1 dose of ABT-335 plus a statin in the preceding double-blind studies or preceding open-label year 1 study, and in this open-label year 2 study. Only subjects with a combination therapy baseline value and postbaseline value at Week 104 are included.
Measure: Median (Full Range); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 162 | 43 | 80
percent change | -36.9 (34.91) [-84.8 to 124.4] | -29.6 (36.61) [-73.1 to 53.0] | -38.7 (32.31) [-80.8 to 80.2]

3. Secondary Outcome: Mean Percent Change in High-Density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 HDL-C minus baseline HDL-C)/baseline HDL-C] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 162 | 43 | 80
percent change | 13.7 (22.15) | 11.2 (22.53) | 5.2 (17.53)

4. Secondary Outcome: Mean Percent Change in Direct Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 LDL-C minus baseline LDL-C)/baseline LDL-C] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 161 | 43 | 80
percent change | -19.2 (30.87) | -20.2 (22.56) | -20.5 (30.04)

5. Secondary Outcome: Mean Percent Change in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 Non-HDL-C minus baseline Non-HDL-C)/baseline Non-HDL-C] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 162 | 43 | 80
percent change | -26.9 (26.12) | -23.8 (21.99) | -25.1 (27.83)

6. Secondary Outcome: Mean Percent Change in Very Low-Density Lipoprotein Cholesterol (VLDL-C) From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 VLDL-C minus baseline VLDL-C)/baseline VLDL-C] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 158 | 42 | 79
percent change | -33.7 (42.50) | -18.7 (58.37) | -26.6 (65.88)

7. Secondary Outcome: Mean Percent Change in Total Cholesterol (Total-C) From Baseline to Week 104 of This Open-Label Year 2 Study
Description: [(Week 104 Total-C minus baseline Total-C)/baseline Total-C] X 100. Baseline is the last value prior to the first dose of combination therapy.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Number analyzed (Participants) | 162 | 43 | 80
percent change | -20.1 (21.41) | -17.9 (18.54) | -20.4 (21.57)

ADVERSE EVENTS:
Time Frame: Up to 116 weeks
Description: Anytime after initiation of combination therapy (in the preceding 12-week double-blind studies or in the preceding open-label year 1 study) to within 30 days after the last dose of combination therapy.
Arm/Group | ABT-335 + 20 mg Rosuvastatin | ABT-335 + 40 mg Simvastatin | ABT-335 + 40 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 26/174 | 4/50 | 5/86
Other Adverse Events (participants affected / at risk) | 153/174 | 44/50 | 81/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + 20 mg Rosuvastatin (N=174) | ABT-335 + 40 mg Simvastatin (N=50) | ABT-335 + 40 mg Atorvastatin (N=86)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-335 + 20 mg Rosuvastatin (N=174) | ABT-335 + 40 mg Simvastatin (N=50) | ABT-335 + 40 mg Atorvastatin (N=86)
Anaemia (Blood and lymphatic system disorders) | 9 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 2
Constipation (Gastrointestinal disorders) | 10 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 14 | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 4 | 4
Nausea (Gastrointestinal disorders) | 18 | 6 | 10
Toothache (Gastrointestinal disorders) | 10 | 1 | 3
Vomiting (Gastrointestinal disorders) | 9 | 3 | 4
Chest discomfort (General disorders) | 1 | 3 | 1
Fatigue (General disorders) | 12 | 4 | 5
Oedema peripheral (General disorders) | 2 | 0 | 7
Pain (General disorders) | 11 | 3 | 5
Pyrexia (General disorders) | 5 | 0 | 6
Seasonal allergy (Immune system disorders) | 2 | 1 | 5
Bronchitis (Infections and infestations) | 24 | 8 | 20
Gastroenteritis (Infections and infestations) | 10 | 3 | 6
Gastroenteritis viral (Infections and infestations) | 5 | 1 | 5
Influenza (Infections and infestations) | 8 | 4 | 11
Nasopharyngitis (Infections and infestations) | 27 | 7 | 10
Sinusitis (Infections and infestations) | 24 | 5 | 10
Upper respiratory tract infection (Infections and infestations) | 49 | 17 | 24
Urinary tract infection (Infections and infestations) | 19 | 3 | 5
Viral infection (Infections and infestations) | 3 | 3 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 5 | 5 | 3
Blood creatine phosphokinase increased (Investigations) | 9 | 4 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 6 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 7 | 15
Bursitis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 7 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 6 | 10
Dizziness (Nervous system disorders) | 15 | 6 | 5
Headache (Nervous system disorders) | 37 | 12 | 20
Paraesthesia (Nervous system disorders) | 7 | 3 | 1
Depression (Psychiatric disorders) | 6 | 3 | 5
Insomnia (Psychiatric disorders) | 16 | 2 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 1
Hypertension (Vascular disorders) | 12 | 3 | 4

LIMITATIONS AND CAVEATS:
This was an open-label study designed to assess the long-term safety of the combination therapies. Evaluation of efficacy outcomes was a secondary objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Provide ABBOTT at least sixty (60) days prior to submission for review, ABBOTT shall return comments within sixty (60) days of receipt of draft. Proposed draft shall be delayed an additional sixty (60) days in addition to the Review Period.